CLINICAL TRIAL: NCT04324593
Title: Healthy Volunteer Study to Evaluate the Impact of Various Common Interventions on Venous Pressure Signal Captured by Peripheral Intravenous Analysis (PIVA) Technology
Brief Title: Healthy Volunteer Study to Evaluate the Impact of Various Common Interventions on Venous Pressure Signal Captured by PIVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to COVID-19
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BXU544319; Pro00041143 (Other: Advarra)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- IV line with an attached Deltran BP transducer (Experimental): After device setup, subjects will be guided through a series of manipulations of the IV set while waveforms, pulse rate (PR), respiratory rate (RR) are collected at the start and stop of each test. At the end of the study, the PIVA algorithm will then be applied to the waveforms and calculated values will be compared with those from bedside monitors to understand the effect of common manipulations on the waveforms and determine most optimal conditions for capturing RR and PR through peripheral IV analysis.
  Interventions: Device: Peripheral intravenous analysis (PIVA) algorithm

INTERVENTIONS:
Device: Peripheral intravenous analysis (PIVA) algorithm — An IV line with an attached Deltran BP transducer will be used together with LabChart software to record venous waveforms during various interventions. These waveforms will be processed using the PIVA algorithm and the calculated values will be compared to those from Nellcor respiratory monitor, Capnograph and cardiac telemetry monitoring.

SUMMARY:
Non-invasive sensors have been used in research in the United States (US) to aid in the assessment of a subject's heart rate (HR), respiratory rate (RR) and fluid volume status. This estimate and its trended value over time, when used along with clinical signs and symptoms and other subject test results, can aid in the process of reaching a diagnosis and formulating a therapeutic plan when abnormalities of volume status, or RR are suspected.

Non-invasive sensors like the Peripheral IntraVenous Analysis (PIVA) sensor under development by Baxter and the Deltran blood pressure (BP) transducer, capture waveforms created by physiological mechanisms such as blood flow and breathing. An algorithm is then applied to the captured waveform to give clinicians an idea of hemodynamic (volume) status, and RR.

In this study, the functional robustness (e.g., subjects sitting, elevated leg positions, etc.) of the PIVA algorithm/technology will be demonstrated by evaluating the impact of various common interventions on the venous pressure signal. All subjects will undergo 33 interventions expected to take approximately 4 - 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Has reviewed, understood and signed an informed consent.
* Age between 18-55 years.
* Body mass index between 18.5-35 kg/m2 with a minimum weight of 45 kg.
* Willing and able to comply with study procedures and duration.
* Subjects wearing any type of nail polish and/or acrylic nails must be willing to remove them prior to admission.

Exclusion Criteria:

* Female subjects who are pregnant.
* Subjects who are currently participating in, or have within the past 30 days participated in, another interventional clinical study or have used an investigational device or drug within the past 30 days.
* Subjects with known respiratory conditions including but not limited to:

  * uncontrolled / severe asthma
  * flu / influenza
  * pneumonia / bronchitis
  * shortness of breath / respiratory distress
  * respiratory or lung surgery
  * emphysema, chronic obstructive pulmonary disease, lung disease
  * any other health condition that the Principal Investigator thinks can affect respiratory health
* Subjects with self-reported heart or cardiovascular conditions including but not limited to:

  * hypertension
  * history of cardiovascular surgery
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * restrictive or constrictive cardiomyopathy
  * congenital heart disease other than patent foramen ovale, repaired atrial or ventricular septal defect
  * any type of cardiac valve disease
  * history of cardiac arrhythmias
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes
  * uncontrolled thyroid disease
  * kidney disease / chronic renal impairment
  * history of seizures (except childhood febrile seizures)
  * epilepsy
  * history of unexplained syncope
  * history of migraine attacks in the last 3 months
  * head injury within the last 2 months
  * cancer / chemotherapy
  * other known health condition should be considered upon disclosure in health assessment form
  * history of substance abuse or addiction to alcohol and or drugs within the last 12 months
* Subjects with self-reported bleeding disorders including but not limited to:

  * hemophilia
  * von Willebrand disease
  * history of blood clots
  * history of bleeding problems
  * bruises easily with everyday activities
* Subjects taking prescription blood thinners (like aspirin, clopidogrel, dipyridamole, or ticlopidine).
* Subjects may be excluded at the discretion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Signal Quality Index (SQI) Score by Supine, Sitting, Standing Body Positions | End of interventions #15 (supine for 5 minutes), #17 (sitting for 5 minutes), and #19 (standing for 5 minutes)
  Ranking of subject body positions (supine, sitting, standing) based upon their impact on the venous waveform signal, from best to worst, based on the PIVA algorithm-derived SQI. Score on the scale include 0=no signal, 1=poor signal, 2=good signal. The highest percentage of time with good signal quality will be the best ranked position, and the lowest percentage of time with good signal quality will be the worst ranked position.

SECONDARY OUTCOMES:
Agreement between PIVA algorithm-derived RR and RR measured with Capnography at Baseline | End of 10 minute baseline
  The difference of the PIVA algorithm-derived outcomes to their comparators (Capnography) under different conditions will be summarized descriptively by n, mean, median, minimum, and maximum. The 95% limit of agreement and a Bland Altman plot will also be done for these endpoints. Capnography is the monitoring of the concentration or partial pressure of carbon dioxide in the respiratory gases.
Agreement between PIVA algorithm-derived RR and RR measured with Nellcor bedside monitor at Baseline | End of 10 minute baseline
  The difference of the PIVA algorithm-derived outcomes to their comparators (Nellcor) under different conditions will be summarized descriptively by n, mean, median, minimum, and maximum. The 95% limit of agreement and a Bland Altman plot will also be done for these endpoints.
Agreement between PIVA algorithm-derived RR and RR measured with manual counting | End of 10 minute baseline
  The manual count value will be an average of the 2 minutes then the count is taken over. The difference of the PIVA algorithm-derived outcomes to their comparators (manual) under different conditions will be summarized descriptively by n, mean, median, minimum, and maximum. The 95% limit of agreement and a Bland Altman plot will also be done for these endpoints.
Agreement between PIVA algorithm derived PR and PR measured with Nellcor bedside monitor at Baseline | End of 10 minute baseline
  The difference of the PIVA algorithm-derived outcomes to their comparators (Nellcor) under different conditions will be summarized descriptively by n, mean, median, minimum, and maximum. The 95% limit of agreement and a Bland Altman plot will also be done for these endpoints.
Change in PIVA algorithm derived volume index between supine and passive leg raising positions | End of Interventions #15 (supine for 5 minutes) and #18 (passive leg raise for 5 minutes)
  The change in PIVA algorithm-derived volume index for a change in positions will be summarized descriptively by n, mean, median, minimum, and maximum.
Change in PIVA algorithm derived volume index between supine and standing positions | End of interventions #15 (supine for 5 minutes) and #19 (standing for 5 minutes)
  The change in PIVA algorithm-derived volume index for a change in positions will be summarized descriptively by n, mean, median, minimum, and maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No